CLINICAL TRIAL: NCT03632486
Title: Bedside Ultrasound Predicts Progression of Severity of Disease in Dengue Fever
Status: Completed | Type: Observational
Sponsor: Timothy Gleeson (Other)
Collaborators: Angkor Hospital for Children (Other)
Responsible Party: Sponsor-Investigator, Timothy Gleeson, Assistant Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: H00003325
Record Dates: First submitted 2018-07-10; First posted 2018-08-15 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Dengue; Fever
Keywords: Ultrasound; Dengue
MeSH Terms: conditions — Dengue; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Dengue: Children with fever and two of the following criteria: anorexia and nausea, rash, aches and pains, warning signs, leukopenia, positive tourniquet test will all receive a diagnostic bedside ultrasound.
  Interventions: Other: Bedside Ultrasound

INTERVENTIONS:
Other: Bedside Ultrasound — Patients enrolled in this study will undergo bedside ultrasound during their initial presentation to the emergency department. Ultrasound imaging protocols include the following:
  * FAST Exam - Standard images will be obtained using the abdominal transducer. Images include the following: 1) sub-xyphoid 2)right upper quadrant (with right thorax) 3)left upper quadrant (with left thorax) and 4) suprapubic
  * Right Upper Quadrant Exam - Standard images will be obtained using the abdominal transducer. Images include the following: 1) Long axis of the gallbladder 2) Transverse axis of the gallbladder fundus 3) Transverse axis of the gallbladder body and 4) Transverse axis of the gallbladder neck.
  * Lung ultrasound to assess for pleural effusions and sonographic b lines.

SUMMARY:
The purpose of this study is determine the ability of bedside ultrasound performed in the Emergency Department and Outpatient Department can predict the severity of disease during a Dengue Fever outbreak in children, in Siem Reap, Cambodia. Our hypothesis is that the presence of gallbladder wall thickening, pulmonary edema/effusions, ascites, pericardial effusion in children correlates with progression to more severe disease.

DETAILED DESCRIPTION:
Dengue fever has various levels of severity, from mild disease to severe hemorrhagic complications and shock. Dengue is endemic world-wide and has been found in the United States. The mortality from dengue fever can be as high as 15-20%, with nearly 22,000 deaths annually, most of them children (Reddy, 2013). There is no reliable way to immediately predict which children presenting with a fever during a Dengue fever outbreak will progress to more severe disease. Some children with dengue fever will improve with limited clinical interventions, but others require intensive therapy. Limited healthcare resources in developing countries make decisions on treatment or disposition difficult as many children and poor clinical decision increase morbidity and mortality. In more developed countries such as the United States, early identification of patients with dengue fever has the potential to identify children who may benefit from early interventions. Identifying those patients is the first step in exploring early therapies to effect mortality. Previous research has demonstrated that intrathoracic/ peritoneal fluid and gallbladder wall thickening is associated with more severe disease for hospitalized patients with dengue (Michels, 2013). The investigators will explore earlier presentations to the emergency department and outpatient department.

The study hypothesis is that the presence of early sonographic findings in children correlates with progression to more severe disease. The study specific aim is to determine the association between sonographic features of dengue and disease progression and clinical outcome in children with dengue fever.

This study is a prospective observational clinical study in the emergency department of the Angkor Hospital for Children in Siem Reap, Cambodia. Study subjects will include children 16 years or less, who present during a dengue outbreak with suspected dengue. Subjects include children with an acute febrile illness and criteria for dengue based on 2010 WHO guidelines (fever and two of the following criteria: anorexia and nausea, rash, aches and pains, warning signs, leukopenia, positive tourniquet test). Clinicians will determine their clinical suspicion of dengue, intended therapeutic interventions and disposition following a history and physical exam. Study personnel will perform diagnostic bedside ultrasound imaging of the gallbladder, peritoneal, cardiac, and pleural spaces. Patients will be followed to determine clinical outcome, therapeutic interventions and disposition. The primary endpoint is progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Fever
2. Clinical suspicion of non-severe dengue (with or without warning signs). (WHO 2010 guidelines)
3. Not a prisoner or ward of the state
4. Parents able and willing to give consent.

Exclusion Criteria:

* Allergic to US gel
* Known pleural or pericardial effusion
* Unstable vital signs
* Severe dengue

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study subjects will include children 16 years or less, who present during the annual dengue outbreak with suspected dengue fever. Subjects include children with fever and two of the following criteria: anorexia and nausea, rash, aches and pains, warning signs, leukopenia, positive tourniquet test.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical Progression of disease | 10 days
  Follow up of Patients to determine hospitalization or treatement

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD PhD, Principal Investigator — UMass Worcester
Locations (1):
- Angkor Hospital for Children, Siem Reap, Cambodia

IPD SHARING:
Plan to Share IPD: No